CLINICAL TRIAL: NCT07300514
Title: Golidocitinib Versus Placebo as Maintenance Therapy for Peripheral T-Cell Lymphoma in Complete or Partial Remission After First-Line Chemotherapy: A Multicenter, Randomized, Double-Blind Phase III Clinical Study.
Brief Title: Golidocitinib Versus Placebo as Maintenance Therapy for Peripheral T-Cell Lymphoma
Acronym: T-START-M1
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T-START-M1-2025
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T-Cell Lymphoma (PTCL NOS); Anaplastic Large Cell Lymphoma, ALK-Negative; Angioimmunoblastic T-cell Lymphoma (AITL); T-follicular Helper Phenotype Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma; ALK-positive anaplastic large cell lymphoma; Angioimmunoblastic T-cell lymphoma; TFH phenotype PTCL; Golidocitinib; JAK1 inhibitor; Maintenance therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to golidocitinib or placebo as maintenance therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind treatment; golidocitinib and placebo are identical in appearance. Tumor assessments are evaluated by investigators and a blinded independent central review (BICR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Experimental: Golidocitinib (Experimental): Participants receive golidocitinib 150 mg orally every other day in 28-day cycles for up to 24 months, or until disease progression, unacceptable toxicity, start of new anti-lymphoma therapy, withdrawal of consent, or study termination.
  Interventions: Device: PET-CTandct- DNAdetection
- Arm B - Placebo Comparator: Placebo (Placebo Comparator): Participants receive matching placebo capsules orally every other day in 28-day cycles for up to 24 months, or until disease progression, unacceptable toxicity, start of new anti-lymphoma therapy, withdrawal of consent, or study termination.
  Interventions: Device: PET-CTandct- DNAdetection

INTERVENTIONS:
Device: PET-CTandct- DNAdetection — The patients who achieved CMR by PET-CT and MRD-neg by ct-DNA testing were evaluated at 12 months,One patient stopped maintenance treatment, while the rest continued for one year.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III trial evaluating golidocitinib as maintenance therapy in adult patients with peripheral T-cell lymphoma (PTCL) who achieved complete response (CR) or partial response (PR) after first-line systemic chemotherapy and are not candidates for hematopoietic stem cell transplantation (HSCT) or decline HSCT. Eligible patients with histologically confirmed PTCL subtypes (PTCL-NOS, ALK-positive anaplastic large cell lymphoma [ALK-ALCL], angioimmunoblastic T-cell lymphoma [AITL], or follicular helper T-cell phenotype PTCL [FTCL/PTCL-TFH]) according to the 2016 WHO classification will be randomized 1:1 to receive oral golidocitinib or matching placebo.

Study treatment is given at 150 mg every other day in 28-day cycles for up to 2 years or until disease progression, unacceptable toxicity, start of new anti-lymphoma therapy, withdrawal of consent, or study termination. At 12 months, patients who achieve complete metabolic response on PET-CT and minimal residual disease (MRD)-negative status by ctDNA may discontinue maintenance, whereas others continue treatment up to 24 months. After treatment discontinuation, patients will be followed for disease status and survival for up to approximately 13 additional cycles. The primary endpoint is progression-free survival (PFS) assessed by investigators per Lugano 2014 criteria. Key secondary endpoints include overall survival, response rates, duration of response, time to next anti-lymphoma therapy, MRD dynamics by ctDNA, and safety.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) are aggressive non-Hodgkin lymphomas with poor prognosis and high relapse rates after first-line chemotherapy. There is no established standard of care for post-remission maintenance therapy in patients who are not candidates for hematopoietic stem cell transplantation. Aberrant activation of the JAK/STAT pathway plays a critical role in the pathogenesis and progression of PTCL. Golidocitinib (Chinese name: 戈利昔替尼) is an oral, potent, and highly selective JAK1 inhibitor that has demonstrated robust antitumor activity and a favorable safety profile in relapsed or refractory PTCL in prior clinical studies, leading to its recommended phase II dose of 150 mg once daily.

Based on these data and the unmet need for effective maintenance strategies, this phase III study (T-START-M1) will enroll adult patients with histologically confirmed PTCL subtypes (PTCL-NOS excluding primary cutaneous disease, ALK-ALCL, AITL, FTCL/PTCL-TFH) who achieved CR or PR after first-line CHOP, BV-CHP, or CHOP-like regimens and are ineligible for HSCT (age >65 years) or decline HSCT despite eligibility. Randomization (1:1) will be stratified by initial response status (CR vs PR), histologic subtype (ALK-ALCL vs others), and HSCT eligibility (ineligible vs eligible-but-declining).

Participants will receive golidocitinib 150 mg every other day or matching placebo in 28-day cycles for up to 24 months. Tumor response will be assessed by imaging according to Lugano 2014 criteria, and ctDNA-based MRD will be evaluated at baseline, 12 months, and end of treatment. Patients who achieve complete metabolic response plus MRD negativity at 12 months may stop maintenance, while others continue up to 2 years. After treatment discontinuation, patients will be followed for progression, subsequent anti-lymphoma therapies, and survival for up to approximately 13 additional cycles (about 1 year). The primary objective is to determine whether golidocitinib maintenance improves PFS compared with placebo. Key secondary objectives include evaluation of overall survival, complete response rate, duration of response, time to next anti-lymphoma therapy, ctDNA-based MRD dynamics, and safety including incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and grade ≥3 AEs.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to any study-specific procedures and willingness to comply with all study requirements.
* Age ≥18 years at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 without deterioration within 2 weeks before screening.
* Histologically confirmed PTCL according to the 2016 WHO classification, limited to the following subtypes: PTCL-not otherwise specified (excluding primary cutaneous PTCL), ALK-positive anaplastic large cell lymphoma (ALK-ALCL), angioimmunoblastic T-cell lymphoma (AITL), or T-follicular helper phenotype PTCL (FTCL or PTCL-TFH).
* Achieved complete response (CR) or partial response (PR) after first-line systemic standard chemotherapy with CHOP, BV-CHP, or CHOP-like regimens, as assessed by Lugano 2014 criteria; patients must be ineligible for HSCT (age >65 years) or eligible but decline HSCT (age ≤65 years). The interval between completion of first-line therapy and planned first dose in this study must be ≤3 months.
* Adequate bone marrow and organ function, including:

  * Absolute neutrophil count (ANC) ≥1.5×10⁹/L (≥1.0×10⁹/L if bone marrow is involved by lymphoma), without use of colony-stimulating factors within 7 days before study entry.
  * Platelet count ≥100×10⁹/L (≥75×10⁹/L if bone marrow is involved by lymphoma), without transfusion or platelet growth factors within 7 days before study entry.
  * Hemoglobin ≥10 g/dL.
  * Total bilirubin ≤2× upper limit of normal (ULN).
  * ALT and AST ≤2.5×ULN.
  * Serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (calculated or measured).
  * Left ventricular ejection fraction (LVEF) ≥50% on echocardiography.
  * Willingness and ability to comply with study procedures and follow-up.

Exclusion Criteria:

* Ann Arbor stage I disease at initial diagnosis.
* Prior treatments that could interfere with study therapy, including but not limited to:

  * Investigational agents or antineoplastic drugs within 30 days before first study dose.
  * Cytotoxic chemotherapy within 21 days before first study dose.
  * Systemic corticosteroids at a prednisone-equivalent dose >10 mg/day within 7 days before first study dose.
  * Major surgery (excluding vascular access procedures) or severe trauma within 4 weeks before first study dose, or planned surgery during study treatment.
  * Antineoplastic monoclonal antibodies (including brentuximab vedotin) within 4 weeks before first study dose; radiotherapy within 3 weeks; other toxin- or radioisotope-conjugated antibodies within 10 weeks.
  * Prior treatment with any JAK or STAT3 inhibitor.
  * Antitumor immunotherapy (e.g., immune checkpoint inhibitors including PD-1, PD-L1, CTLA-4 antibodies) within 28 days before first study dose.
  * Live attenuated or viral vector vaccines within 28 days before first study dose.
  * Current use of vitamin K antagonists, antiplatelet or anticoagulant drugs that cannot be discontinued ≥7 days before first study dose.
  * Concomitant medications that are strong CYP3A inducers or inhibitors, or BCRP/P-gp substrates with narrow therapeutic index that cannot be stopped ≥7 days before first study dose, as specified in the protocol appendix.
* Active hepatitis C infection (positive anti-HCV antibody).
* Hepatitis B virus (HBV) DNA ≥1000 IU/mL or other HBV status not meeting protocol-defined criteria for safe inclusion.
* Known HIV infection with confirmed positive serology.
* Any uncontrolled, clinically significant comorbidities or laboratory abnormalities that, in the investigator's judgment, would increase risk or interfere with study participation.
* History of drug-induced interstitial lung disease or current evidence of clinically significant interstitial lung disease.
* Pregnant or breastfeeding women; women of childbearing potential and men with fertile partners who are unwilling or unable to use effective contraception during treatment and for the protocol-specified period after the last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From randomization to the first documentation of disease progression, relapse, or death from any cause, up to approximately 3 years.
  PFS is defined as the time from randomization to the first documented disease progression or relapse according to Lugano 2014 criteria, or death from any cause, whichever occurs first, as assessed by investigators. A blinded independent central review (BICR) will perform a sensitivity analysis of PFS to assess robustness.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death from any cause, up to approximately 5 years.
  Time from randomization to death from any cause.
Complete Response Rate (CRR) | From randomization to end of treatment, up to 24 months.
  Proportion of patients achieving complete response (CR) according to Lugano 2014 criteria.
Duration of Response (DOR) | From the first documented response (CR or PR) to disease progression, relapse, or death, up to approximately 3 years.
  Duration of response among patients who achieve CR or PR.
Time to Next Anti-lymphoma Therapy (TTNT) | From randomization to the start of the next systemic anti-lymphoma therapy or death, up to approximately 3 years.
  ime from randomization to the first administration of subsequent anti-lymphoma therapy or death.
MRD Negativity Rate by ctDNA at 12 Months | 12 months after randomization.
  Proportion of patients who achieve minimal residual disease (MRD)-negative status by ctDNA assessment at 12 months.
Incidence of Treatment-emergent Adverse Events (TEAEs) | From first dose of study drug to 28 days after the last dose.
  Number and percentage of patients experiencing TEAEs, serious adverse events (SAEs), grade ≥3 AEs, AEs leading to dose interruption, dose reduction, or treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD &PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellei M, Foss FM, Shustov AR, Horwitz SM, Marcheselli L, Kim WS, Cabrera ME, Dlouhy I, Nagler A, Advani RH, Pesce EA, Ko YH, Martinez V, Montoto S, Chiattone C, Moskowitz A, Spina M, Biasoli I, Manni M, Federico M; International T-cell Project Network. The outcome of peripheral T-cell lymphoma patients failing first-line therapy: a report from the prospective, International T-Cell Project. Haematologica. 2018 Jul;103(7):1191-1197. doi: 10.3324/haematol.2017.186577. Epub 2018 Mar 29. PMID 29599200
- [Result] Maurer MJ, Ellin F, Srour L, Jerkeman M, Bennani NN, Connors JM, Slack GW, Smedby KE, Ansell SM, Link BK, Cerhan JR, Relander T, Savage KJ, Feldman AL. International Assessment of Event-Free Survival at 24 Months and Subsequent Survival in Peripheral T-Cell Lymphoma. J Clin Oncol. 2017 Dec 20;35(36):4019-4026. doi: 10.1200/JCO.2017.73.8195. Epub 2017 Oct 26. PMID 29072976
- [Result] Park SI, Horwitz SM, Foss FM, Pinter-Brown LC, Carson KR, Rosen ST, Pro B, Hsi ED, Federico M, Gisselbrecht C, Schwartz M, Bellm LA, Acosta M, Advani RH, Feldman T, Lechowicz MJ, Smith SM, Lansigan F, Tulpule A, Craig MD, Greer JP, Kahl BS, Leach JW, Morganstein N, Casulo C, Shustov AR; COMPLETE Investigators. The role of autologous stem cell transplantation in patients with nodal peripheral T-cell lymphomas in first complete remission: Report from COMPLETE, a prospective, multicenter cohort study. Cancer. 2019 May 1;125(9):1507-1517. doi: 10.1002/cncr.31861. Epub 2019 Jan 29. PMID 30694529
- [Result] Maurer B, Nivarthi H, Wingelhofer B, Pham HTT, Schlederer M, Suske T, Grausenburger R, Schiefer AI, Prchal-Murphy M, Chen D, Winkler S, Merkel O, Kornauth C, Hofbauer M, Hochgatterer B, Hoermann G, Hoelbl-Kovacic A, Prochazkova J, Lobello C, Cumaraswamy AA, Latzka J, Kitzwogerer M, Chott A, Janikova A, Pospisilova S, Loizou JI, Kubicek S, Valent P, Kolbe T, Grebien F, Kenner L, Gunning PT, Kralovics R, Herling M, Muller M, Rulicke T, Sexl V, Moriggl R. High activation of STAT5A drives peripheral T-cell lymphoma and leukemia. Haematologica. 2020 Jan 31;105(2):435-447. doi: 10.3324/haematol.2019.216986. Print 2020. PMID 31123029
- [Result] Cooley L, Dendle C, Wolf J, Teh BW, Chen SC, Boutlis C, Thursky KA. Consensus guidelines for diagnosis, prophylaxis and management of Pneumocystis jirovecii pneumonia in patients with haematological and solid malignancies, 2014. Intern Med J. 2014 Dec;44(12b):1350-63. doi: 10.1111/imj.12599. PMID 25482745
- [Result] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Result] Armitage JO. The aggressive peripheral T-cell lymphomas: 2017. Am J Hematol. 2017 Jul;92(7):706-715. doi: 10.1002/ajh.24791. PMID 28516671